CLINICAL TRIAL: NCT05130450
Title: An Open-Label Extension Study of AKCEA-APOCIII-LRx Administered Subcutaneously to Patients With Familial Chylomicronemia Syndrome (FCS)
Brief Title: A Study of Olezarsen (Formerly Known as AKCEA-APOCIII-LRx) in Participants With Familial Chylomicronemia Syndrome (FCS)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 678354-CS13; 2021-003280-95 (EudraCT Number)
Expanded Access: NCT06360237 (Approved for marketing)
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Familial Chylomicronemia Syndrome
Keywords: FCS
MeSH Terms: conditions — Familial hyperchylomicronemia syndrome | interventions — olezarsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Olezarsen (Experimental): Olezarsen will be administered once every 4 weeks by subcutaneous (SC) injection from Week 1 through Week 153.
  Interventions: Drug: Olezarsen

INTERVENTIONS:
Drug: Olezarsen — Olezarsen will be administered by SC injection.
  Other Names: ISIS 678354; AKCEA -APOCIII-LRx

SUMMARY:
The purpose of this study is to evaluate the effect of olezarsen (formerly known as AKCEA-APOCIII-LRx) on the percent change in fasting triglycerides (TG) from baseline.

DETAILED DESCRIPTION:
This is a multi-center, open-label extension (OLE) study of up to 60 participants with FCS rolling-over from Study ISIS 678354-CS3 (NCT04568434). Participants will receive olezarsen during a 157-week treatment period, followed by a 13-week post-treatment follow-up period. The length of participation in this study is approximately 201 weeks, which includes an up to 31-day qualification period, a 157-week treatment period, and a 13-week post-treatment evaluation period.

Treatment has been extended to obtain additional safety assessments and efficacy data and to provide patients with continued access to ISIS 678354 until the drug may be available commercially.

ELIGIBILITY:
Inclusion Criteria:

• Satisfactory completion of treatment with olezarsen in the index study (ISIS 678354-CS3, last dose as scheduled at Week 49) with an acceptable safety profile, per Investigator judgement.

Exclusion Criteria:

• Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the participant unsuitable for enrollment, or could interfere with the patient participating in or completing the study, including need for treatment with medications disallowed in the index study (ISIS 678354-CS3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in Fasting TG at 6 Months (Average of Weeks 23, 25, and 27) Compared to Baseline | Baseline and 6 months

SECONDARY OUTCOMES:
Percent Change From Baseline in Fasting TG at 12 Months (Average of Weeks 51 and 53) at 24 Months (Average of Week 103 and Week 105) and 36 Months (Average of Week 155 and Week 157) | Baseline and 36 months
Percentage of Participants Who Achieve ≥ 40% Reduction in Fasting TG From Baseline at 6 Months | At 6 months
Percentage of Participants Who Achieve ≥ 40% Reduction in Fasting TG From Baseline at 12, 24, 36 Months | At 12, 24, 36 months
Percent Change in Fasting apoC-III from Baseline at Month 6 | Baseline and 6 months
Percent Change in Fasting apoC-III from Month 12, 24, 36 | At 12, 24, 36 months
Percent Change From Baseline in Fasting Apolipoprotein 48 (apoB48) at 6 Months | At 6 months
Percent Change From Baseline in Fasting apoB48 at 12, 24, 36 Months | At 12, 24, 36 months
Percent Change in Fasting non-HDL-C from Baseline at Month 6 | Baseline and 6 months
Percent Change in Fasting non-HDL-C from Months 12, 24, 36 | At 12, 24, 36 months
Percentage of Participants Who Achieve Fasting TG ≤ 880 milligrams per deciliter (mg/dL) at 6 Months | At 6 months
Percentage of Participants Who Achieve Fasting TG ≤ 880 mg/dL at 12, 24, 36 months | At 12, 24, 36 months
Adjudicated Acute Pancreatitis Event Rate During the Treatment Period in Participants With ≥ 2 Events of Adjudicated Acute Pancreatitis in 5 Years Prior to Treatment With Study Drug in the Index Study | Week 1 through Week 157
Adjudicated Acute Pancreatitis Event Rate During the Treatment Period | Week 1 through Weeks 53, 105, or 157
Adjudicated Acute Pancreatitis Event Rate During the Treatment Period in Patients with a Prior History of Pancreatitis within 10 Years Prior to Screening in the Index Study | Week 1 through Weeks 53, 105, or 157
Percentage of Participants Who Achieve ≥ 70% Reduction in Fasting TG From Baseline at 6 Months | At 6 months
Percentage of Participants Who Achieve ≥ 70% Reduction in Fasting TG From Baseline at 12, 24, 36 Months | At 12, 24, 36 months
Percentage of Participants Who Achieve Fasting TG ≤ 500 mg/dL at 6 Months | At 6 months
Percentage of Participants Who Achieve Fasting TG ≤ 500 mg/dL at 12, 24, 36 Months | At 12, 24, 36 months

CONTACTS AND LOCATIONS:
Locations (27):
- United States (7):
  - Diabetes/Lipid Management & Research Center, Huntington Beach, California
  - Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - Department of Pharmacy, Park Ridge, Illinois
  - University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - CTSI Investigational Pharmacy, New York, New York
  - Milstein Hospital, New York, New York
  - IDS Central, Philadelphia, Pennsylvania
- Canada (4):
  - Ecogene-21, Chicoutimi, Quebec
  - Institute de Recherches Cliniques de Montreal, Montreal, Quebec
  - Nathalie Saint-Pierre, Montreal, Quebec
  - Clinique des Maladies Lipidiques de Quebec Inc., Québec, Quebec
- France (3):
  - Groupement Hospitalier Est- Pharmacie Secteur Essais Clinique, Bron
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Pharmacie Hopital de la Conception, Marseille
- Italy (3):
  - Via Sergio Pansini 5, Napoli
  - UOC di Farmacia AOUP PAOLO GIACCONE, Palermo
  - Azienda Ospedaliero Universitaria Policlinico Umberto I, Rome
- Academisch Medisch Centrum Goederenontvangst Apotheek t.a.v. Kenniscentrum, Amsterdam, Noor-Holland, Netherlands
- Oslo Hospital Pharmacy Rikshospitalet, Oslo, Norway
- Portugal (2):
  - Hospital da Senhora da Oliveira Guimaraes, Creixomil
  - Dra Margarida Falcao Centro Hospitalar Lisboa Ocidental Hospital Egas Moniz, Lisbon
- Metabolicke centrum MU, Bratislava, Slovakia
- Spain (3):
  - Hospital Clínic Barcelona C/ Villarroel, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
- Apokteket AB, Malmo, Sweden
- Royal Manchester Children's Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.
URL: https://vivli.org/ourmember/ionis/